CLINICAL TRIAL: NCT05476276
Title: EPPIC-Net: Platform Protocol to Assess Treatments for Painful Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: James P. Rathmell, MD (Other)
Collaborators: New York University (Other); Icahn School of Medicine at Mount Sinai (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, James P. Rathmell, MD, Chair, Department of Anesthesiology, Perioperative and Pain Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022P002381 (EN21-PP); 5U24NS113850-03 (NIH)
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: The Platform Protocol is intended to potentially accommodate different design plans for different assets. In addition, it is anticipated that the protocol may evolve over time, as lessons learned from earlier assets are used to fine tune the study design for later assets in an adaptive approach. For reasons of generalizability (including consideration of minimizing participant burden and being attractive to asset holders), a parallel-group design will typically be employed, and it is the current intention that designs should provide 80% power to detect an effect size of 0.35 on the primary efficacy outcome
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization assignment within an ISA will be blinded from study participants, staff from clinical sites, investigators, asset owners, IND sponsors, and/or designees. This blinding will be accomplished by providing identical investigational product and packaging for each asset and its corresponding control treatment. The use of IXRS will ensure the blinding is accomplished.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EN21-01 ISA (Experimental): The EN21-01 Intervention Specific Analysis is detailed in the protocol (NCT#)
  Interventions: Drug: ISA specific
- Placebo Comparator (Placebo Comparator): Each ISA will detail the use of the Placebo Comparator.
  Interventions: Drug: ISA specific

INTERVENTIONS:
Drug: ISA specific — ISA specific interventions will be listed in their protocols.

SUMMARY:
This is a Platform Protocol to perform Phase II clinical trials in The Early Phase Pain Investigation Clinical Network (EPPIC-Net), under The Helping to End Addiction Long-termSM Initiative, or NIH HEAL InitiativeSM, related to the treatment of Painful Diabetic Peripheral Neuropathy (PDPN) in a platform setting to test multiple assets under a single protocol.

DETAILED DESCRIPTION:
This is a Platform Protocol that allows evaluation of more than one treatment in a single trial structure, to be run within EPPIC-Net. Instead of testing individual assets in a series of clinical trials, this Platform Protocol sets out the framework for testing multiple assets related to PDPN. This provides an efficient approach to evaluate multiple therapies under a single infrastructure in a timely fashion. The Platform Protocol also allows efficiencies by creating the possibility of sharing information across assets, such as data from control conditions.

This Platform Protocol is for a platform design to allow for the testing of multiple assets. Some platform trials allow direct comparisons of competing therapies for the same condition. However, for this EPPIC-Net platform trial, there will not be direct comparisons of assets to one another. Instead, assets will only be compared to a placebo. This is in service to the EPPIC-Net primary goal of accelerating the development of pain treatment because, based on feedback from asset-holders, the possibility of comparison of assets to one another or to an active drug would be a deterrent for asset-holders' participation in EPPIC-Net.

ELIGIBILITY:
3.1. Platform Protocol Inclusion Criteria (To be used in conjunction with ISA-specific criteria. Note, some ISA criteria may be more stringent than Platform criteria; always follow the more stringent criteria when determining eligibility.)

Participants must meet all of the following inclusion criteria:

1. Able to provide informed consent. Legally Authorized Representatives (LARs) are not allowed, but impartial witnesses may be utilized as needed for visually impaired participants.
2. 18 years of age and older
3. Diagnosis of diabetes mellitus
4. Meets the Toronto Criteria for probable clinical sensorimotor polyneuropathy, with PDPN symptoms present for at least six months. This is defined as a combination of symptoms and signs with any two or more of the following (must be present bilaterally in the distal lower extremities): neuropathic symptoms, decreased distal sensation, or unequivocally decreased (or absent) ankle reflexes. Specifically:

   1. The presence of any neuropathic symptoms on either the "Douleur Neuropathique en 4 Questions" (DN4) or the EPPIC-Net Neuropathy Exam will suffice to demonstrate "neuropathic symptoms."
   2. Decreased distal sensation is satisfied by any of the following:

   i. "Yes" is checked at least once under Question 3 of the DN4 which queries hypoesthesia to touch and pinprick.

   ii. At least one score of "reduced" or "absent" on the right AND at least one score of "reduced" or "absent" on the left in any of the following items from the EPPIC-Net Neuropathy Exam:
   * Pin sensation in segments 1 or 2 (i.e. the toes and feet)
   * Vibration at the great toe
   * Joint position at the great toe
   * Light touch/touch pressure at the great toe
   * Temperature at the great toe
   * Monofilament at the great toe c. Decreased or absent ankle reflexes is satisfied by a score of "reduced" or "absent" on the right AND left in the "Ankle reflex" item in the EPPIC-Net Neuropathy Exam.
5. A score of at least 4 on the "Douleur Neuropathique en 4 Questions" (DN4).
6. Pain reporting during a pre-defined 7-day screening period meets study criteria (to be established using a centrally-administered screening algorithm) which may account for mean pain intensity reported, variability in reported values, and adherence in reporting.
7. Patient reported daily 11-point NRS (for average and worst pain over the last 24 hours) is completed on at least 5 out of the 7 days in the screening and baseline periods.
8. Participants must be willing and able to comply with scheduled visits, the treatment schedule, laboratory testing, and other requirements of the study (e.g., completion of app-based daily reporting).
9. Females may be included if they meet at least one of the following criteria (note that individual ISAs may specify more stringent measures to prevent pregnancy):

   a. Are not of childbearing potential, defined as one or more of the following: i. Post-menopausal for at least 1 year ii. Surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) iii. XY genotype iv. Turner syndrome v. Uterine agenesis. b. Are completely abstinent from sexual activity capable of resulting in pregnancy (as part of their preferred and usual lifestyle). This will include females whose sole sexual partner is a male who has undergone surgical sterilization or vasectomy.

   c. Women of childbearing potential will agree to practice an effective form of two types of birth control, which are defined as those, alone or in combination, that result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. This must be done before, throughout, and for 30 days after the last dose of DB study drug. Acceptable methods are: i. Hormonal methods such as the vaginal ring, or oral, implantable, injectable, or transdermal contraceptives for a minimum of 1 full cycle (based on the participant's usual menstrual cycle period) before study drug administration.

   ii. Intrauterine device. iii. Barrier method of contraception: condoms with or without a spermicidal agent, diaphragm or cervical cap with spermicide
10. Specific requirements of male participants (regarding contraception) will be defined in the ISAs based on the potential toxicity profile of the asset.

3.2. Platform Protocol Exclusion Criteria (To be used in conjunction with ISA-specific criteria; note, some ISA criteria may be more stringent than Platform criteria; always follow the more stringent criteria when determining eligibility)

Please note that some of the below criteria which depend on clinical judgment require contacting the MM. Participants must not meet any of the following exclusion criteria, organized by category:

3.2.1. Neuropathy Confound Exclusion Criteria

1. Peripheral neuropathy that is known to have been caused by a condition other than diabetes (e.g. HIV, cancer/chemotherapy-induced, other medication-induced, alcohol-induced, hereditary, autoimmune neuropathies, uncontrolled or untreated hypothyroidism). Note that participants will not be tested for HIV, this will be established by patient report or review of the medical record.
2. Other significant pain conditions involving the same area as the neuropathy (e.g. physical deformity of the feet, plantar fasciitis, lumbosacral radiculopathy with distal lower extremity pain, fibromyalgia involving the lower limbs, Morton's neuroma), that in the opinion of the investigator would interfere with the participant's ability to rate the neuropathy pain.
3. Other pain conditions not involving the same area as the neuropathy which (in the opinion of the investigator) interfere with the participant's ability to rate the neuropathy pain.
4. Any amputation of the lower limb which interferes with the participant's ability to rate the neuropathy pain. If there is any amputation please contact the MM to confirm eligibility prior to randomization to an ISA.
5. The presence of any current foot ulcer.
6. Significant peripheral vascular disease defined as symptoms consistent with intermittent claudication.

   3.2.2. Medication/Treatment Exclusion Criteria
7. Use of other investigational drugs within 3 months before screening and throughout the study.
8. Known or suspected hypersensitivity to all of the assets (active component and excipients) currently being tested in the Platform Protocol.
9. Undergone neurolytic or neurosurgical therapy or used an implanted neurostimulating device for neuropathic pain in the distal lower limbs within 3 months of screening.
10. Use of the high dose capsaicin patch (8%) in the 6 months before screening and throughout the study (for the treatment of PDPN). Use of the capsaicin patch in a manner that is not expected to interfere with the measurement of PDPN severity is allowed.
11. Participants who meet any of the following regarding concomitant treatments:

    1. Unwilling or unable to discontinue episodic or periodic treatments for pain in the distal legs and/or feet (e.g., injections of local anesthetics).
    2. Starting a new non-pharmacological pain treatment (e.g. relaxation/hypnosis, physical or occupational therapy, any exercise-based therapy, any talk-based therapy, acupuncture, TENS) for the treatment of PDPN within 4 weeks prior to screening OR planning on starting a new non-pharmacologic treatment for PDPN OR planned changes to a stable non-pharmacologic treatment for PDPN during the study.

    i. Non-pharmacological treatment for conditions other than PDPN is allowed without restriction.
12. Active use of opioids or marijuana for any reason at screening and unwilling or unable to discontinue use.

    3.2.3. Medical Exclusion Criteria
13. Clinically significant ECG or laboratory abnormalities at the Screening Visit that would put the participant at undue risk or affect the ability of the participant to participate in the trial (in the opinion of the investigator). Screening ECG and lab results may be repeated without requiring a rescreen, as long as the participant is still within the screening window.
14. Participants whose glycemic control has been unstable within 3 months before screening (e.g. ketoacidosis requiring hospitalization).
15. Proliferative retinopathy or maculopathy requiring acute treatment.
16. Requiring dialysis.
17. Myocardial infarction or stroke in the past 6 months.
18. Known diagnosis of moderate to severe hepatic impairment (equivalent to Child-Pugh class B or C) OR aspartate aminotransferase or alanine aminotransferase ≥ 3 times the upper limit of normal during the screening process.
19. A clinically significant illness or operative procedure within 4 weeks of screening.
20. Clinically significant surgery planned during the study period. If a surgery is planned, please contact the MM for approval before randomization.
21. History of malignancy or other medical condition that would put the participant at undue risk or affect the ability of the participant to participate in the trial (in the opinion of the investigator).
22. Pregnant or nursing. 3.2.4. Psychosocial and Substance Use Disorders Exclusion Criteria
23. A clinically significant psychiatric disease that would put the participant at undue risk or affect the ability of the participant to participate in the trial (in the opinion of the investigator).
24. Alcohol use disorder or other substance use disorders (other than nicotine or caffeine) in accordance with DSM-5 criteria within 12 months of screening.
25. Positive urine drug tests defined as one or more of the following (see Urine Drug Testing Section 6.2.13.5.1):

    1. Two positive urine drug tests for a prescribed opioid (buprenorphine, opiates, methadone and/or oxycodone), prior to the initiation of investigational product (IP);
    2. Two positive urine drug tests for marijuana (prescribed or recreational), prior to the initiation of investigational product (IP);
    3. One positive urine drug test for cocaine, ecstasy, methamphetamines, or phencyclidine (PCP);
    4. One positive urine drug test for non-prescribed amphetamines, barbiturates, benzodiazepines, or opioids (buprenorphine, opiates, methadone and/or oxycodone).
26. Vulnerable persons defined as either of the following:

    1. Individuals whose willingness to volunteer in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of a retaliatory response from senior members of a hierarchy in case of refusal to participate.

Individuals whose judgment has been impaired by their physical, mental, or socio-economical condition and those incapable of giving informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Daily 0-10 pain NRS | Past 24 hours
  Typically, the primary efficacy endpoint for this Platform Protocol will be based on the daily 0-10 pain NRS. Participants will respond to the following every evening before going to bed:
  * "Select the number that best describes your average neuropathy pain during the past 24 hours."
  * "Select the number that best describes your worst neuropathy pain during the past 24 hours."
  Typically, the primary efficacy endpoint for this Platform Protocol will be based on the daily 0-10 pain NRS. Participants will respond to the following every evening before going to bed:
  * "Select the number that best describes your average neuropathy pain during the past 24 hours."
  * "Select the number that best describes your worst neuropathy pain during the past 24 hours."

SECONDARY OUTCOMES:
Pain, Enjoyment, and General activity scale (PEG) | Past 24 hours
  The PEG is a three-item (each scored 0-10) multidimensional pain measure designed and validated for use in primary care and other ambulatory clinic patients, as a practical and useful tool to improve assessment and monitoring of chronic pain in primary care.
Pain Catastrophizing Scale - Short Form 6 (PCS-SF6) | Past 24 hours
  Catastrophizing is a pain-specific psychosocial construct comprising cognitive and emotional processes such as helplessness, pessimism, rumination about pain-related symptoms, and magnification of pain reports. The PCS-SF6 is a 6-item, self-report measure of catastrophic thinking associated with pain. Scores range from 0-24, with higher scores indicating more catastrophizing.
PROMIS Physical Functioning Short-Form 6b | Past 24 hours
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Functioning short form is a 6-item scale that is widely used in pain research. It is a unidimensional scale that shows broad coverage of the physical function construct, good construct validity, and high levels of temporal stability. The PROMIS Physical Function Scale is expressed as a T-score, with a population mean of 50 and SD of 10. Higher scores represent better physical functioning; possible T scores in this distribution range from 21 to 59 (PROMIS, 2020).
Pain Health Questionnaire (PHQ-2) | Past 24 hours
  The 2-item PHQ-2 is a brief depression screening tool that correlates strongly with PHQ-9 scores and shows good sensitivity for identifying individuals with depressive disorders in the general population in a variety of medical samples. Scores range from 0-6, with higher scores indicating more depressive symptomatology.
Generalized Anxiety Disorder - 2 item scale (GAD-2) | Past 24 hours
  The GAD-2 is a 2-item screening tool that is widely used to screen for clinically significant anxiety symptoms and anxiety disorders in clinical settings. It shows good sensitivity and specificity as a screening tool for anxiety disorders. Scores range from 0-6, with higher scores indicating more anxiety symptomatology.
Patient Global Impression of Change (PGIC) | Past 24 hours
  The PGIC is a single-item measure of patient-reported improvement that is widely used as a general outcome measure in studies of chronic pain patients. It is often used as an index of treatment-associated change, and patient-reported improvements in the form of PGIC scores correlate robustly with significant improvement in pain intensity, pain interference with activities of daily living, mood, and quality of life (Perrot and Lanteri-Minet, 2019).
Tobacco, Alcohol, Prescription medication, and other Substance use Tool (TAPS-1) | Past 24 hours
  The TAPS-1 is the screening component of the TAPS tool and consists of a single stem question with four items covering the frequency of past-12-month use of tobacco, alcohol, and illicit drugs, and non-medical use of prescription medications. Scores range from 0-4; higher scores indicate a higher likelihood of problematic substance use. The TAPS-1 shows good sensitivity and specificity for identifying substance use disorders.
PROMIS Sleep Disturbance - 6A | Past 24 hours
  The PROMIS Sleep Disturbance short form is a convenient 6-item scale that correlates strongly with the longer forms. The PROMIS Sleep Disturbance Scale is expressed as a T-score, with a population mean of 50 and standard deviation (SD) of 10. Possible T scores in this distribution range from 31.7 to 76.1 (PROMIS, 2021).
Sleep Duration | Past 24 hours
  A single-item scale measuring the duration of actual sleep a participant has gotten, on average, over the past month. Numerical responses will be provided in hours and minutes.
Opioid Use Questionnaire (OUQ) | Past 24 hours
  The OUQ is an indicator of past or present use of any of the listed opioid medications. There are a total of three yes/no items where a yes indicates the use of such medications

OTHER OUTCOMES:
Norfolk Quality of Life - Diabetic Neuropathy (Norfolk QOL-DN) | Past 24 hours
  The Norfolk QOL-DN is a validated 47-item, patient-reported outcome measure, sensitive to the different features of diabetic neuropathy (DN) including small fiber, large fiber, and autonomic function.
Neuropathy Examination | Past 24 hours
  The neuropathy examination will be a single consolidated procedure consisting of visual inspection of the feet, brief distal motor exam, ankle and knee deep tendon reflexes, and a standardized sensory exam. This single exam will collect all the data needed to calculate several common scores including: the Michigan Neuropathy Screening Instrument (MNSI) Part B (Feldman et al., 1994; Herman et al., 2012), the Utah Early Neuropathy Scale (UENS) (Singleton et al., 2008), and the Toronto Clinical Scoring System (Toronto CSS) (Bril & Perkins, 2002). Disambiguation: Toronto CSS is the name given to the scale initially. In a subsequent publication (Bril et al, 2008) this scale is referred to as the Toronto Clinical Neuropathy Score (TCNS), and its modification as the modified Toronto Clinical Neuropathy Score (mTCNS).

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Robinson-Papp, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (23):
- United States (23):
  - University of California, San Diego, San Diego, California
  - South Lake Pain Institute, Clermont, Florida
  - SIMEDHealth LLC, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Northwestern Department of Neurology, Chicago, Illinois
  - Healthcare Research Network (Flossmoor), Flossmoor, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland - Baltimore, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - MGH Department of Anesthesia, Critical Care, and Pain, Boston, Massachusetts
  - Healthcare Research Network (Hazelwood), Hazelwood, Missouri
  - Columbia University Medical Center/Neurological Institute, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester, Rochester, New York
  - Clinical Inquest Center, Beavercreek, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Low Country Pain Center, Orangeburg, South Carolina
  - Nerve and Muscle Center of Texas, Houston, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - VCU Department of Neurology, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
The use of Global Unique Identifiers (GUIDs) allows data to be linked with a given research participant, without revealing any of the participant's identifiable information. All participants in NIH-funded research must have a GUID. This study is using the Biomedical Research Informatics Computing System (BRICS) GUID platform to assign GUIDs. This ID should be generated at the time of Informed Consent since it requires several pieces of patient information (e.g., last name at birth, first name at birth, sex at birth, day, month and year of birth, city and country of birth, etc.). The GUID will be a combination of letters and numbers to form a unique identifier, e.g. TBIAC412JJK. Sites should maintain a list to link the GUID to the participant.